CLINICAL TRIAL: NCT03402867
Title: Effects of Myofascial Trigger Point Dry Needling on Neck Pain in Orchestral Musicians
Brief Title: Effects of Dry Needling on Neck and Shoulder Pain in Orchestral Musicians: a Prospective Case Series
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CEU San Pablo University (Other)
Responsible Party: Principal Investigator, Aitor Martin-Pintado Zugasti, PhD, CEU San Pablo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEU-012
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Pain Syndrome; Musculoskeletal Pain; Trigger Point Pain, Myofascial
MeSH Terms: conditions — Somatoform Disorders; Musculoskeletal Pain; Myofascial Pain Syndromes

STUDY DESIGN:
Intervention Model Description: Deep dry needling
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Deep dry needling applied on active myofascial trigger points in the shoulder and neck regions
  Interventions: Procedure: Deep dry needling

INTERVENTIONS:
Procedure: Deep dry needling — Insertion of a filiform needle in the active trigger point of musculoskeletal muscle

SUMMARY:
This study evaluates the effectiveness of Deep dry needling of active myofascial trigger points present in muscles of the neck and shoulder region in orchestral musicians.

ELIGIBILITY:
Inclusion Criteria:

* Orchestral musicians
* Chronic neck or shoulder pain
* Presence of active myofascial trigger points

Exclusion Criteria:

* Fear of needles
* Coagulation disorders
* Pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale for pain | 2 weeks
  Pain measurement. 100-mm visual analog scale (VAS), horizontal line ranging from 0mm (no pain) to 100mm (worst imaginable pain).

SECONDARY OUTCOMES:
Pressure pain threshold | 2 weeks
  Analogic algometer
Neck disability index (NDI) | 2 weeks
  10-item, 50-point index that assesses different aspects of daily functioning in patients with neck pain. It assesses four items regarding subjective symptoms (pain intensity, headache, concentration, sleeping), four items regarding activities of daily living (lifting, work, driving, recreation), and two items regarding discretionary activities of daily living (personal care, reading). Each item is scored 0 to 5, with the total reported as either a raw score (0-50) or as a percentage score. Higher values represent a worse outcome.
Shoulder pain disability index (SPADI) | 2 weeks
  Self-administered questionnaire, grouping 13 questions, 5 of which measure the severity of pain caused by various arm movements involving the shoulder, the pain being assessed on a numeric pain scale ranging from 0 to 10. Eight additional questions related to functional impairments of the shoulder are assessed with a numeric scale. Higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- CEU San Pablo University, Madrid, Madrid, Spain